CLINICAL TRIAL: NCT06628583
Title: Multivariate Analysis and Risk Factors Were Used to Predict the Short-term Postoperative Pain of Degenerative Lumbar Spine
Status: Completed | Type: Observational
Sponsor: Hao Liu (Other)
Responsible Party: Sponsor-Investigator, Hao Liu, Chief orthopaedic surgeon, First Affiliated Hospital of Suzhou University, China, First Affiliated Hospital of Suzhou Medical College
Organization: First Affiliated Hospital of Suzhou Medical College (Other)
Other Study IDs: (2024) Lun Yan Grant No. 518
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Disc Herniation; Lumbar Degenerative Disease; Sarcopenia
Keywords: Lumbar Degenerative disease; PLIF; Sarcopenia; Sagittal bit balance; Machine learning
MeSH Terms: conditions — Intervertebral Disc Displacement; Sarcopenia | interventions — Magnetic Resonance Spectroscopy; Contrast Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The study did not involve biological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rehabilitation Group: mild/non pain group with VAS<3 at 3th months after PLIF.N=501
  Interventions: Other: Magnetic Resonance Imaging with Contrast
- Recurrent pain group: Recurrent pain group: recurrent pain group with VAS≥3 at 3th months after PLIF.N=435
  Interventions: Other: Magnetic Resonance Imaging with Contrast

INTERVENTIONS:
Other: Magnetic Resonance Imaging with Contrast — The study was retrospective and did not set interventions

SUMMARY:
The objective of this retrospective clinical study wasto study the risk factors for short-term low back and leg pain after PLIF in patients with lumbar Degenerative disease, and to establish a risk prediction model for short-term low back and leg pain after PLIF based on relevant risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of lumbar degenerative disease (spinal stenosis, disc herniation with lumbar instability, and lumbar spondylolisthesis), with no significant symptomatic relief after conservative treatment for more than 3 months, and in need of surgical intervention;
2. lumbar spinal fusion surgical treatment with PLIF;
3. grouping based on the presence or absence of a lumbar or limb pain with VAS ≥3 at the 3th month postoperative follow-up;
4. observational indicators including individual factors, surgical factors, spine-pelvis sagittal balance parameters, and paravertebral muscle parameters.

Exclusion Criteria:

(1) those with a history of lumbar spine trauma, inflammation, tumor, or surgery; (2) those with congenital or acquired severe lumbar vertebral deformity; (3) those with severe neurological dysfunction; (4) those with incomplete baseline and follow-up data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The data of 936 patients who underwent PLIF for lumbar Degenerative disease from June 2018 to March 2023 were collected retrospectively. The patients were divided into rehabilitation group（N=501） and residual pain group（N=435）according to their postoperative pain
Sampling Method: Non-Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
General situation of the patient | Before the operation
  General information such as age, sex, BMI and psychological status was collected

SECONDARY OUTCOMES:
Surgical situation | 1-3 months after surgery
  It includes the course of disease, the operation time, the amount of bone cement injected during the operation, the leakage of bone cement and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Medical record system and imaging system of the First Affiliated Hospital of Suzhou University, China, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes